CLINICAL TRIAL: NCT00005624
Title: A Multicenter Phase 2 Study of Oral N-Acetyl Dinaline (CI-994) in the Treatment of Patients With Advanced Myeloma
Brief Title: CI-994 in Treating Patients With Advanced Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Parke-Davis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-11560; PD-994-04 (Other: Parke-Davis); NCI-G00-1758 (Other: NCI)
Record Dates: First submitted 2000-05-02; First posted 2004-07-26 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Multiple Myeloma
Keywords: refractory multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; plasma cell neoplasm
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — tacedinaline; Histone Deacetylase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CI-994 Treatment (Experimental): Patients receive CI-994 orally daily. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed for 30 days and then every 2 months.
  Interventions: Drug: CI-994

INTERVENTIONS:
Drug: CI-994 — CI-994 as outlined in treatment arm.
  Other Names: Oral N-Acetyl Dinaline; Tacedinaline; HDAC Inhibitor; CAS 112522-64-2; Acetyldinaline; PD 123654

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of CI-994 in treating patients who have advanced myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the antitumor activity of CI-994 in patients with advanced myeloma. II. Determine the response rate, response duration, and overall survival of this patient population with this treatment regimen. III. Determine the safety of this treatment in these patients.

OUTLINE: This is a multicenter study. Patients receive CI-994 orally daily. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed for 30 days and then every 2 months.

PROJECTED ACCRUAL: A total of 8-63 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage IIA or IIIA myeloma with a measurable M- component in the serum or urine Progressing disease after conventional chemotherapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Greater than 8 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 75,000/mm3 (transfusion independent) Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) AST/ALT no greater than 2 times ULN Renal: Creatinine no greater than 1.5 times ULN Calcium no greater than 12 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception No life threatening illness unrelated to the tumor No concurrent serious infection No prior malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix Must be capable of swallowing intact medication capsules No medical or psychiatric condition that would prevent written informed consent

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 14 days since prior immunologic agents No concurrent immunologic agents Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy No concurrent chemotherapy Endocrine therapy: At least 2 weeks since prior high dose corticosteroids No concurrent anticancer hormonal therapy No concurrent corticosteroids Radiotherapy: At least 3 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 1997-08; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 5 years
  Response Rate according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria.

SECONDARY OUTCOMES:
Duration of Response | 5 years
  Response of duration in months
Number of Participants with Overall Survival (OS) | 5 years
  Participants surviving at end of study.
Number of Participants with Adverse Events | 5 years
  Review of adverse events utilizing Common Toxicity Criteria (CTC) V3.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Alsina, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States